CLINICAL TRIAL: NCT03361800
Title: A Non-randomized, Non-comparative, Open-label, Window Trial of Entinostat Given With or Without Exemestane in Patients With Newly Diagnosed, Stage I-IIIC, Hormone Receptor - Positive (HR+) or Triple Negative Breast Cancer (TNBC)
Brief Title: Window of Opportunity Trial of Entinostat in Patients With Newly Diagnosed Stage I-IIIC,TNBC
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Funding withdrawn.
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Syndax Pharmaceuticals (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: LCCC 1639; P50CA058223 (NIH)
Record Dates: First submitted 2017-11-28; First posted 2017-12-05 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Breast Cancer; Invasive Breast Cancer; ER-Negative PR-Negative HER2-Negative Breast Cancer
Keywords: Breast Cancer; ER Negative Breast Cancer; Triple Negative Breast Cancer; PR Negative Breast Cancer; ER Positive PR Positive Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — entinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Entinostat (Experimental): Nine days prior to their scheduled surgery, entinostat 5mg PO given once weekly on day 1 and day 8
  Interventions: Drug: Entinostat

INTERVENTIONS:
Drug: Entinostat — oral drug, 5mg tablet given once weekly x 2 doses

SUMMARY:
This study is investigational and is not designed to treat cancer. In other words, the study drug, entinostat, is not being given to treat cancer. Instead, the study team is looking at the effects of entinostat on tumor tissue for research purposes only.

Approximately 246,660 cases of breast cancer were diagnosed in the United States in 2016. Its detection and treatment remains a major concern in women's healthcare. In particular, TNBC accounts for approximately 15-20% of all breast cancers. Research into treatment for breast cancer relies more and more on understanding how the cancer cells act when they are exposed to an anti-cancer drug. How most cancer cells act when exposed to anti-cancer drugs and which patients as a result may benefit the most from these drugs is not well known. Additional studies are required to determine the cells' reactions. The purpose of part 1 of this study is to better understand how TNBC tumors react to one particular cancer drug, entinostat. Entinostat is currently being studied across multiple clinical trials for the treatment of breast cancer, other solid tumors and blood cancers. Entinostat is investigational and has not yet been FDA approved for the treatment of cancer.

Studies have shown that a good way to determine how cancer acts when exposed to anti-cancer drugs is a short-term preoperative window study. In this type of study, subjects receive a study drug a couple of days before surgery. Leftover tissue from surgery is then used to determine some of the effects that a study drug may have on the tumor. In this study, subjects will receive two doses of entinostat prior to undergoing planned surgery. Leftover tissue from this surgery will then be used to determine the effects entinostat has on tumor cells. For example, the study team will examine if the types of genes and proteins that the tumor expresses as a result of entinostat exposure increases or decreases the likelihood that the tumor will not continue to grow. A gene is a unit of DNA. Genes make up the chemical structure carrying your genetic information that may determine human characteristics (i.e., eye color, height and sex). This study will focus on discovering how entinostat affects a wide variety of genes in tumor cells.

DETAILED DESCRIPTION:
Primary Objective and Endpoint To identify decrease in Ki-67 mRNA following treatment with entinostat across TNBC breast cancers.

Secondary Objectives and Endpoints To identify messenger ribonucleic acid (mRNA) gene expression changes following treatment with entinostat, across TNBC.

To evaluate changes in the proliferation signature by mRNA expression following treatment with entinostat across TNBC.

To identify differential kinome activation before and after treatment with entinostat across TNBC

To correlate mutation and/or copy number variations by whole exome sequencing (WES) with mRNA gene expression changes and reduction of proliferation signature following treatment with entinostat across TNBC.

To correlate protein lysine hyperacetylation in peripheral blood and tumor from pre- and post-entinostat treated TNBCs.

To explore molecular subtype, Programmed death-ligand 1 (PD-L1) and other immune checkpoint molecule expression, immune gene and innate anti-programed cell death-1 resistance (IPRES) expression signatures and phenotypes of tumor-infiltrating lymphocytes, including delineation of effector and regulatory T cells, and define T cell receptor (TCR) repertoire prior to and following entinostat treatment in TNBCs. We will also explore mutation and copy number variation status, and predicted major histocompatibility complex (MHC) class I neoantigen burden.

To document safety of entinostat in patients with TNBC prior to their scheduled surgical resection per National Cancer Institute - Common Terminology for Adverse Events (NCI-CTCAE v4.0).

ELIGIBILITY:
Inclusion Criteria:

* Is female, age ≥ 18 years of age.
* For Part 1: Has histologically confirmed newly diagnosed Stage I-IIIC invasive breast cancer that is triple negative (ER/PR <1%, Her2 negative) and is scheduled to undergo definitive surgery (either lumpectomy, mastectomy) and meets the criteria listed below:

  1. Scheduled for lumpectomy or mastectomy and not considered a candidate for neoadjuvant systemic treatment
  2. No prior or current therapy for breast cancer
  3. Amenable to a baseline research breast biopsy

For Part 2: Has histologically confirmed newly diagnosed Stage I-IIIC invasive breast cancer that is ER positive (+/- PR positive) and is scheduled to undergo definitive surgery (either lumpectomy, mastectomy) and meets the criteria listed below:

* Scheduled for lumpectomy or mastectomy and not considered a candidate for neoadjuvant systemic treatment b. No prior or current therapy for breast cancer c. Amenable to a baseline research breast biopsy
* Must have sufficient time to receive two doses of entinostat 7 days apart or exemestane for 8 consecutive days with or without entinostat prior to surgery.
* Has an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1.
* Demonstrates adequate organ function
* Has normal cardiac function based on an electrocardiogram (ECG) with no clinically significant abnormalities or risks including any of the following:

  * Current uncontrolled hypertension (systolic >150 mm Hg and/or diastolic >100 mmHg) or unstable angina
  * History of serious cardiac arrhythmia requiring treatment (exceptions: atrial fibrillation, paroxysmal supraventricular tachycardia)
  * History of myocardial infarction within 6 months of day 1 of dosing
  * History of congestive heart failure according to New York Heart Association (NYHA) criteria.
* For women of childbearing potential: Has a negative serum pregnancy test at screening within 72 hrs of receiving study treatment. In addition, female subjects must either:

  1. agree to the use of an approved method of contraception (ie, two adequate barrier methods throughout the study starting with the screening visit) and to continue its use for the duration of the study treatment through 120 days after the last dose of entinostat if a woman of child-bearing potential, or
  2. has documented inability to become pregnant (e.g., hysterectomy, bilateral tubal ligation or oophorectomy, or post-menopausal as defined as total cessation of menses for ≥ 2 years). Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound. Tubal ligation must be confirmed with medical records of the actual procedure otherwise the patient must be willing to use 2 adequate barrier methods throughout the study.
* Is able to swallow and retain oral medication.
* As determined by the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures for the entire length of the study.

Exclusion Criteria:

* Stage IV breast cancer.
* Has clinically significant a) abnormal laboratory or ECG findings, b) history of myocardial infarction or arterial thromboembolic events within 6 months of screening or c) unstable angina, d) New York Heart Association (NYHA) Class III or IV disease or e) a corrected QT (QTc) interval > 470 msec.
* Medical history of uncontrolled hypertension (NCI CTCAE grade 3 or 4) or diabetes mellitus.
* Known active central nervous system metastases and/or carcinomatous meningitis.
* Prior history of another cancer within the previous 5 years with the exception of adequately treated basal cell carcinoma or cervical intraepithelial neoplasia, cervical carcinoma in situ or melanoma in situ.
* Another known malignancy other than breast cancer that is progressing or requires active treatment.
* Is pregnant or lactating, or is of child-bearing potential and not willing to use an approved method of contraception.
* Has a concomitant medical condition that precludes adequate study treatment compliance or assessment, such as bleeding disorders or any other medical condition that would increase risks of additional core biopsy for biomarkers.
* Is currently receiving treatment with a medication on the prohibited medication list for entinostat (See section 11.1 Appendix A and section 4.5).
* Has allergy to benzamides or inactive components of the study medication (entinostat).
* Inability to take oral medications (eg, impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral medications such as ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection).
* Is participating in another therapeutic clinical trial or has received another investigational agent within 30 days prior to informed consent.
* Known human immunodeficiency virus (HIV), Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV) infection (with the exception of chronic or cleared HBV and HCV infection which is allowed).
* Has acute or currently active/requiring anti-viral therapy, hepatic or biliary disease (with the exception of patients with Gilbert's syndrome, asymptomatic gallstones, or stable chronic liver disease per investigator assessment).
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study.
* Medical history of an autoimmune disease that requires ongoing steroid therapy for > 14 days.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-11-28 (Actual); Primary Completion 2019-09-18 (Actual); Study Completion 2019-10-11 (Actual)

PRIMARY OUTCOMES:
Decrease in Ki-67 mRNA following treatment with entinostat across TNBC breast cancers | 9 days from start of entinostat (day of surgery)
  RNA will be extracted from tumor samples using the Qiagen RNEasy Mini RNA extraction kit. mRNA-Seq libraries will made according to the Illumina TruSeq RNA Access protocol. Determination of molecular subtypes and relative expression of genes (i.e. Ki-67 as primary objective) and gene signatures from mRNA-seq data will be done. Change (decrease) in Ki-67 mRNA expression from will be measured by log2 fold-change in Ki-67 mRNA-seq expression from pre-treatment to post-treatment within each patient.

SECONDARY OUTCOMES:
mRNA gene expression changes following treatment with entinostat, across TNBC | 9 days from start of entinostat (day of surgery)
  RNA will be extracted from tumor samples using the Qiagen RNEasy Mini RNA extraction kit. mRNA-Seq libraries will made according to the Illumina TruSeq RNA Access protocol. Determination of molecular subtypes and relative expression of genes (i.e. Ki-67 as primary objective) and gene signatures from mRNA-seq data will be done. Expression of mRNA-seq will be measured in terms of relative standard error of the mean (RSEM) expected read counts after normalization by upper quartile normalization to adjust for between-sample differences in library sizes.
Changes in the proliferation signature by mRNA expression following treatment with entinostat across TNBC | 9 days from start of entinostat (day of surgery)
  RNA will be extracted from tumor samples using the Qiagen RNEasy Mini RNA extraction kit. mRNA-Seq libraries will made according to the Illumina TruSeq RNA Access protocol. Determination of molecular subtypes and relative expression of genes (i.e. Ki-67 as primary objective) and gene signatures from mRNA-seq data will be done. Genes belonging to the proliferation signature will be individually examined and summarized by descriptive statistics.
Differential kinome activation before and after treatment with entinostat across TNBC | 9 days from start of entinostat (day of surgery)
  Tissue samples for pre-treatment kinome analysis will be obtained from tissue remaining from the diagnostic, pre-treatment baseline biopsy (or from additional core needle biopsy of accessible tissue at study entry, if insufficient tissue is available from the diagnostic biopsy). Tissue samples for post-treatment kinome analysis will be obtained from the surgical procedure. A chemical proteomics approach will be employed to define the activity of a significant percentage of the expressed kinome in cells and tumors. Differential kinome activation will be measured in terms of the log2 fold change in MaxQuant Label Free Quantification (LFQ) intensity before and after treatment.
Correlation of mutation and/or copy number variations by whole exome sequencing (WES) with mRNA gene expression changes and reduction of proliferation signature following treatment with entinostat across TNBC. | 9 days from start of entinostat (day of surgery)
  The T-cell receptor (TCR) repertoires of tumors and matched peripheral blood samples pre and post treatment with entinostat will be profiled, as well as the presence of dominant tumor-infiltrating clonotypes in the peripheral blood. RNA and whole-exome sequencing on tumor samples will be performed to capture molecular subtype, PD-L1 and other immune checkpoint molecule expression, immune gene signature and IPRES expression (ie, IPRES is a transcriptional signature associated with innate anti-PD-1 resistance) mutation and copy number variation status, and predicted MHC class I neoantigen burden. Continuous variables such as mRNA expression and DNA copy number will be assessed via Spearman Correlation, and correlation between categorical variables such as mutations and T-cell Phenotype will be assessed via Fisher's Exact Test.
Correlation of protein lysine hyperacetylation in peripheral blood and tumor from pre- and post-entinostat treated TNBCs | 9 days from start of entinostat (day of surgery)
  Changes in protein lysine acetylation in blood mononuclear cells (PBMCs) will be assessed using an assay developed by the Trepel Laboratory, NCI/NIH. Pre to post-treatment change in protein lysine acetylation.will be measured in terms of the log2 fold change in MaxQuant LFQ intensity before and after treatment, and will be summarized with descriptive statistics
Percentage of participants with treatment related adverse events | 30 days after treatment with entinostat
  Any patient who receives at least one dose of entinostat on this protocol will be evaluable for toxicity, with toxicity evaluated using the National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI CTCAE) v4.0.
  Safety assessments will consist of monitoring and reporting adverse events (AEs) and serious adverse events (SAEs) that are considered related to entinostat, all events of death, and any study specific issue of concern.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Carey, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comprehensive Cancer Center at University of North Carolina, Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No